CLINICAL TRIAL: NCT02595645
Title: GENESIS: Genetic Biopsy for Prediction of Surveillance Intervals After Endoscopic Resection of Colonic Polyps
Acronym: GENESIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Collaborators: Technical University of Munich (Other); Medical University of Graz (Other); Specialized Medical Office for Gastroenterology Dornstadt (Other); QIAGEN Gaithersburg, Inc (Industry)
Responsible Party: Principal Investigator, Thomas Seufferlein, Prof. Dr. Alexander Meining, University of Ulm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: GENESIS
Record Dates: First submitted 2015-10-29; First posted 2015-11-03 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Colonic Polyps
Keywords: colorectal adenoma; colorectal cancer; next generation sequencing; liquid biopsy; screening colonoscopy; surveillance strategies
MeSH Terms: conditions — Colonic Polyps; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Polypectomy and NGS (Experimental): All patients which underwent screening colonoscopy and fulfilling the inclusion criteria are eligible. Polyps were biopsied and underwent histopathological and genetic analyses
  Interventions: Genetic: Polypectomy and NGS

INTERVENTIONS:
Genetic: Polypectomy and NGS — NGS of 38 cancer-related genes, systems biological analyses, correlation genetics to pathology and clinical data

SUMMARY:
Colorectal cancer ist the 2nd most leading cancer among men and women in germany. Screening colonoscopy has the potential to detect premalignant lesions. By endoscopical resection of these lesions, colorectal cancers could be avoided. The decision for surveillance is made according to patients medical history, amount and histological characteristics of the resected polyps. Molecular guided decisions are still missing. Thus, further tools and mechanisms, beyond but in addition to endoscopy and histopathological, are strongly required to reduce such interval carcinomas and get a better and deeper inside into molecular alterations which occurs in premalignant lesions in the colon and describe risk populations which might benefit from shorter surveillance strategies by colonoscopy. Therefore GENESIS will enroll 100 patients, which underwent screening colonoscopy with polyp ectomy. All biopsies were stored and processed without formalin in special boxes (PaxGene by Qiagen®). After microdissection of polyp tissue and isolation of DNA targeted next generation sequencing of 38 cancer-related genes followed by bioinformatics and systems biology analyses. The sequencing results were correlated to the endoscopical and histopathological findings. In parallel we are collecting EDTA-blood samples for analysis of circulating cell-free DNA (cfDNA) to investigate the potential of liquid biopsies in premalignant colorectal lesions.

DETAILED DESCRIPTION:
Colorectal cancer ist the 2nd most leading cancer among men and women in germany. Screening colonoscopy is provided for all people over 55 years in germany to detect and remove precancerous lesions (polyps) and thereby prevent the occurence of colorectal cancers. According to the result of screening colonoscopy and histopathological examination of the removed polyps the next examination will be planned. But so called interval carcinomas were observed with increasing incidence. Thus, further tools and mechanisms, beyond but in addition to endoscopy and histopathology, are strongly required to reduce such interval carcinomas and get a better and deeper inside into molecular alterations which occurs in premalignant lesions in the colon and describe risk populations which might benefit from shorter surveillance strategies by colonoscopy. Therefore we will enroll 100 patients, which underwent screening colonoscopy with polyp ectomy. Each polyp, provided for endoscopical removal, well be biopsied and stored separately. In each case, diagnosis is ensured. Per patient a maximum of 6 biopsies (from 6 different polyps) is intended. All biopsies were stored and processed without formalin in special boxes (PaxGene by Qiagen®). After microdissection of polyp tissue and isolation of DNA targeted next generation sequencing of 38 genes (ACVR1B, DCC, MIER3, SLC9A9, AKT1, DMD, MLH1, SMAD2, APC, EP300, MSH2, SMAD4, ATM, ERBB2, MSH3, TCERG1, ATP6V0D2, FBXW7, MSH6, TCF7L2, BAX, FZD3, MYO1B, TGFBR2, BRAF, GPC6, NRAS, TP53, CASP8, KRAS, PIK3CA, WBSCR17, CDC27, MAP2K4, PIK3R1, CTNNB1, MAP7, PTPN12) followed by bioinformatics and systems biology analyses. The sequencing results were correlated to the endoscopical and histopathological findings. In parallel we are collecting EDTA-blood samples for analysis of circulating cell-free DNA (cfDNA). NGS targeted sequencing of these 38 genes should also be performed on cfDNA level to investigate the potential of liquid biopsies in premalignant colorectal lesions.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* indication of screening colonoscopy

Exclusion Criteria:

* chronic inflammatory bowl disease
* known colorectal cancer (except curative treated colorectal cancers more than 5 years ago)
* disagreement in participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2015-08; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Genetic landscape of colonic polyps based on NGS-analysis | 1 year
  Are we able to describe risk populations based on clinical, histopathological and sequencing data which might bring a benefit for these cohort for shorter surveillance strategies by colonoscopy? What are the similarities in the altered genes, what are the differences? Are we able to define common signaling hubs?

CONTACTS AND LOCATIONS:
Overall Officials: Alexander G. Meining, Prof. Dr., Principal Investigator — University Ulm, Internal Medicine I, Interventional and experimental endoscopy (InExEn)
Locations (4):
- Medical University Graz, Graz, Styria, Austria
- Germany (3):
  - Specialized Medical Office for Gastroenterology, Dornstadt, Baden-Wurttemberg
  - University Ulm, Internal Medicine I, Interventional and Experimental Endoscopy (InExEn), Ulm, Baden-Wurttemberg
  - Technical University Munich, Munich, Bavaria